CLINICAL TRIAL: NCT06223724
Title: Prospective Study of Status Telemetry for Cochlear Implantations
Brief Title: Status Telemetry for Cochlear Implantations
Acronym: PATHOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: PATHOS
Record Dates: First submitted 2023-06-29; First posted 2024-01-25 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cochlear implant electrode insertion depth estimation: Electrode insertion depth estimation using impedance telemetry data measured during cochlear implantation and at three regular follow-up visits
  Interventions: Device: STOP; Device: MAESTRO

INTERVENTIONS:
Device: STOP — Software to measure impedance telemetry data
Device: MAESTRO — Software to measure impedance telemetry data

SUMMARY:
Cochlear implants (CIs) are well-established neuroprosthesis used to restore hearing for patients with partial or complete deafness. However, the audiological outcomes of these implants can vary widely, and one reason for this is suboptimal electrode placement. The gold standard for measuring electrode positions is computed tomography (CT) scans, but they are expensive and expose patients to additional radiation, which is especially harmful for children.

This study investigates an alternative approach using impedance telemetry data to estimate electrode positions without exposing patients to radiation. For this purpose, an extended telemetry version of a CE-certified cochlear implant software is used. The advanced impedance telemetry software can measure impedance subcomponents with improved measurement resolution that could be used for more accurate estimation of electrode insertion depth using specially designed estimation software.

Ultimately, the investigators want to demonstrate the potential to improve audiological outcomes of cochlear implant recipients without exposing them to additional radiation.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Subjects scheduled for CI surgery according to clinical routine
* Subjects who will receive a cochlear implant of the MED-EL portfolio (FLEX series arrays)
* No radiological contraindications
* Stated willingness to comply with all study procedures for the duration of the study

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Subjects incapable of giving informed consent
* Age under 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects eligible for a MED-EL cochlear implant of the MED-EL portfolio (Flex series array) and who meet the additional inclusion/exclusion will be approached for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Linear error of electrode insertion depth estimation | At the first post-operative CT scan according to conventional clinical routine (+0-4weeks)
  Linear error (in mm) in impedance-based estimation of cochlear implant electrode insertion depth compared to ground truth from CT scans.
Linear error of electrode insertion depth estimation | At the additional post-operative CT scan (+3 months)
  Linear error (in mm) in impedance-based estimation of cochlear implant electrode insertion depth compared to ground truth from CT scans.

SECONDARY OUTCOMES:
Intra-operative progression of impedance subcomponents | During cochlear implantation (day 0)
  Intra-operative measurement of access resistance and polarization impedance measured by the STOP software at several positions of the electrode array in the cochlea (stepwise insertion). The results will be expressed in kOhm (kΩ).
Post-operative progression of electrode insertion depth estimation | Recordings will be made during cochlear implant surgery (day 0) and at three follow-up visits (+2weeks, +4weeks, +12weeks).
  Post-operative cochlear implant electrode insertion depth estimation using a phenomenological model based on access resistance and polarization impedance measured by the STOP software after full insertion of the electrode array. The results will be expressed in kOhm (kΩ).
Angular error of electrode insertion depth estimation | At the first post-operative CT scan according to conventional clinical routine (+0-4weeks)
  Angular error (in degrees) in impedance-based estimation of cochlear implant electrode insertion depth using a phenomenological model compared to ground truth from CT scans.
Angular error of electrode insertion depth estimation | At the additional post-operative CT scan (+3 months)
  Angular error (in degrees) in impedance-based estimation of cochlear implant electrode insertion depth using a phenomenological model compared to ground truth from CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Caversaccio, Prof. Dr. med., Principal Investigator — Inselspital, Bern University Hospital Department of ENT, Head and Neck Surgery
Locations (1):
- Inselspital, Bern University Hospital Department of ENT, Head and Neck Surgery, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No